CLINICAL TRIAL: NCT01682434
Title: Wavefront-guided LASIK for Correction of Myopia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institution changed surgical method to small-incision lenticule extraction. Study never started.
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anders Ivarsen, MD, PhD, Aarhus University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AUH_LASIK
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wavefront-guided LASIK (Active Comparator): One eye will be randomized to wavefront-guided treatment. The other receives conventional LASIK.
  Interventions: Procedure: Laser in situ keratomileusis (LASIK)
- Conventional LASIK (Active Comparator): One eye will receive wavefront-guided LASIK. The other eye receives conventional treatment.
  Interventions: Procedure: Laser in situ keratomileusis (LASIK)

INTERVENTIONS:
Procedure: Laser in situ keratomileusis (LASIK) — Wavefront guided treatment in one eye, conventional in the other.
  Other Names: Device: Carl Zeiss Meditec Visumax femtosecond LASIK; Device: Carl Zeiss Meditec MEL-80 excimer laser.

SUMMARY:
Laser in situ keratomileusis is a successful procedure for the treatment of low to moderate myopia.

Advances over the last decade have allowed LASIK to also correct higher order wavefront aberrations. In low myopia, there seem to be a minor effect of such wavefront-guided treatment. However, it remains to be established whether there is a beneficial effect in higher degrees of myopia.

The study aims to determine whether myopic subjects (-6 to -10 diopters) with higher-than-average preoperative higher-order aberrations have benefit of wavefront-guided treatment. Subjects are randomized to wavefront-guided treatment in one eye, and conventional treatment in the other.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 50 years
* No known ocular or systemic disease
* Not pregnant or breastfeeding
* Myopia between -6.0 and -10.0 diopters
* Astigmatism below 2.0 diopters
* Difference of less than 1.0 diopters in spherical equivalent between eyes
* Normal corneal topography
* Corneal thickness sufficient for planned treatment

Exclusion Criteria:

* Patients that do not fulfill inclusion criteria
* Insufficient quality of ocular wavefront measurement

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 months

SECONDARY OUTCOMES:
Ocular higher order aberrations | 12 months
  Hartmann-Schack wavefront aberrometry using the Zeiss Meditec WASCA

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ivarsen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus, Denmark